CLINICAL TRIAL: NCT04571476
Title: Diagnostic Value of Ultrathin and Thin Bronchoscope for Peripheral Pulmonary Lesions: A Prospective Randomized Controlled Multicenter Study
Brief Title: Diagnostic Value of UTB and TB for PPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); West China Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE202002
Record Dates: First submitted 2020-09-26; First posted 2020-10-01 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Pulmonary Lesion
Keywords: Ultrathin bronchoscope; Thin bronchoscope; Peripheral pulmonary lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UTB-VBN-EBUS group (Experimental): Ultrathin bronchoscope with a 3.0-mm outer diameter and a 1.7-mm working channel was used in this group. Specimens were obtained using 1.5-mm biopsy forceps and 1.4-mm cytology brush with the guidance of VBN and EBUS.
  Interventions: Procedure: Ultrathin bronchoscope; Procedure: Virtual bronchoscopic navigation combined with endobronchial ultrasound
- TB-VBN-EBUS-GS group (Active Comparator): Thin bronchoscope with a 4.0-mm outer diameter and a 2.0-mm working channel was used in this group. Specimens were obtained using 1.5-mm biopsy forceps and 1.4-mm cytology brush with the guidance of VBN-EBUS and a 1.95-mm outer diameter guide sheath.
  Interventions: Procedure: Thin bronchoscope; Procedure: Virtual bronchoscopic navigation combined with endobronchial ultrasound; Procedure: Guide sheath
- TB-VBN-EBUS-non-GS group (Active Comparator): Thin bronchoscope with a 4.0-mm outer diameter and a 2.0-mm working channel was used in this group. Specimens were obtained using conventional biopsy forceps and cytology brush with the guidance of VBN and EBUS, but without guide sheath.
  Interventions: Procedure: Thin bronchoscope; Procedure: Virtual bronchoscopic navigation combined with endobronchial ultrasound

INTERVENTIONS:
Procedure: Ultrathin bronchoscope — Ultrathin bronchoscope (UTB) with an outer diameter no more than 3.0-mm and a 1.7-mm working channel.
  Other Names: UTB
  Arms: UTB-VBN-EBUS group
Procedure: Thin bronchoscope — Thin bronchoscope with a 4.0-mm outer diameter and a 2.0-mm working channel.
  Other Names: TB
  Arms: TB-VBN-EBUS-GS group; TB-VBN-EBUS-non-GS group
Procedure: Virtual bronchoscopic navigation combined with endobronchial ultrasound — VBN can create a path to the target lesion automatically when the lesion is depicted in this software.VBN combined with EBUS can improve the diagnostic yield of PPL and shorten the examination time, which has become the standard method for the diagnosis of PPL.
  Other Names: VBN-EBUS
Procedure: Guide sheath — GS is a cannula with the thinnest outer diameter of 1.95 mm.
  Other Names: GS
  Arms: TB-VBN-EBUS-GS group

SUMMARY:
The purpose of the study is to evaluate the diagnostic value and safety of ultrathin and thin bronchoscope (UTB and TB) for peripheral pulmonary lesions (PPLs) without X-ray fluoroscopy.

DETAILED DESCRIPTION:
The study aims to evaluate the diagnostic value and safety of ultrathin and thin bronchoscope (UTB and TB) with the guidance of virtual bronchoscopic navigation (VBN) combined with endobronchial ultrasound (EBUS) for peripheral pulmonary lesions (PPLs) without X-ray fluoroscopy. The study is designed as a prospective, multicenter, randomized controlled clinical trial. The participating centers are The First Affiliated Hospital of Guangzhou Medical University, Cancer Hospital Chinese Academy of Medical Sciences, West China Hospital, Sichuan University, and Henan Provincial People's Hospital. Patients are divided into three groups: UTB-VBN-EBUS group, TB-VBN-EBUS-GS group and TB-VBN-EBUS-non-GS group. Each subject will be randomized to each group. The study is expected to enroll a total of 577 patients with 193, 192 and 192 in UTB-VBN-EBUS group, TB-VBN-EBUS-GS group and TB-VBN-EBUS-non-GS group, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Chest imaging shows the presence of peripheral pulmonary lesions (defined as those lesions that are surrounded by pulmonary parenchyma and located below the segmental bronchus) that need to be confirmed by pathology. The length diameter of the lesion is no less than 8 mm and no more than 5 cm.
* Patients without contraindications of bronchoscopy.
* Patients have good medical adherence and signed informed consent.

Exclusion Criteria:

* Peripheral pulmonary lesion is pure ground-glass opacity.
* Absence of bronchus leading to or adjacent to the lesion on thin-slice chest CT.
* Visible lumen lesions in segment and above segment bronchus during bronchoscopy (evidence of endobronchial lesion, extrinsic compression, submucosal tumor, narrowing, inflammation or bleeding of the bronchus).
* Diffuse pulmonary lesions.
* The investigators believe that patient has other conditions that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | Up to 6 months
  Diagnostic yield of ultrathin and thin bronchoscope for peripheral pulmonary lesions

SECONDARY OUTCOMES:
Total examination time | During the procedure
  Total examination time is defined from the time that the bronchoscope is inserted beyond the glottis, until the bronchoscope has been removed from the glottis after examination
Duration of finding lesions | During the procedure
  Duration of finding lesions defined from insertion of ultrasound probe to withdrawal of ultrasound probe
Feature of lesions | Up to 6 months
  The feature of peripheral pulmonary lesions affecting the diagnostic yield includes the nature, size, location, the position of the ultrasound probe relative to the lesions etc.
Difference in the bronchus level reached with the bronchoscope | During the procedure
  Level: Bronchus is level 0, leaf bronchus is level 1, segment bronchus is level 2, sub-segment bronchus is level 3, and so on, such as: LB3a is level 3
Difference in diagnostic yield | Up to 6 months
  Difference in diagnostic yield between thin bronchoscope with guide sheath combined small biopsy forceps and without guide sheath combined with conventional biopsy forceps.
Complication rate | 1 month
  The complications refer to the total of serious adverse events related to the procedure during or within 1 month after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurimoto N, Miyazawa T, Okimasa S, Maeda A, Oiwa H, Miyazu Y, Murayama M. Endobronchial ultrasonography using a guide sheath increases the ability to diagnose peripheral pulmonary lesions endoscopically. Chest. 2004 Sep;126(3):959-65. doi: 10.1378/chest.126.3.959. PMID 15364779
- [Background] Steinfort DP, Khor YH, Manser RL, Irving LB. Radial probe endobronchial ultrasound for the diagnosis of peripheral lung cancer: systematic review and meta-analysis. Eur Respir J. 2011 Apr;37(4):902-10. doi: 10.1183/09031936.00075310. Epub 2010 Aug 6. PMID 20693253
- [Background] Yoshikawa M, Sukoh N, Yamazaki K, Kanazawa K, Fukumoto S, Harada M, Kikuchi E, Munakata M, Nishimura M, Isobe H. Diagnostic value of endobronchial ultrasonography with a guide sheath for peripheral pulmonary lesions without X-ray fluoroscopy. Chest. 2007 Jun;131(6):1788-93. doi: 10.1378/chest.06-2506. PMID 17565021
- [Background] Asano F, Ishida T, Shinagawa N, Sukoh N, Anzai M, Kanazawa K, Tsuzuku A, Morita S. Virtual bronchoscopic navigation without X-ray fluoroscopy to diagnose peripheral pulmonary lesions: a randomized trial. BMC Pulm Med. 2017 Dec 11;17(1):184. doi: 10.1186/s12890-017-0531-2. PMID 29228929
- [Background] Oki M, Saka H, Asano F, Kitagawa C, Kogure Y, Tsuzuku A, Ando M. Use of an Ultrathin vs Thin Bronchoscope for Peripheral Pulmonary Lesions: A Randomized Trial. Chest. 2019 Nov;156(5):954-964. doi: 10.1016/j.chest.2019.06.038. Epub 2019 Jul 26. PMID 31356810
- [Background] Oki M, Saka H, Ando M, Asano F, Kurimoto N, Morita K, Kitagawa C, Kogure Y, Miyazawa T. Ultrathin Bronchoscopy with Multimodal Devices for Peripheral Pulmonary Lesions. A Randomized Trial. Am J Respir Crit Care Med. 2015 Aug 15;192(4):468-76. doi: 10.1164/rccm.201502-0205OC. PMID 26039792
- [Background] Asano F, Shinagawa N, Ishida T, Shindoh J, Anzai M, Tsuzuku A, Oizumi S, Morita S. Virtual bronchoscopic navigation combined with ultrathin bronchoscopy. A randomized clinical trial. Am J Respir Crit Care Med. 2013 Aug 1;188(3):327-33. doi: 10.1164/rccm.201211-2104OC. PMID 23600452
- [Derived] Feng X, Zhang Q, Luo F, Zhang X, Zhang L, Xie F, Sun J, Li S. Study design for a multicenter, randomized controlled trial evaluating the diagnostic value of ultrathin bronchoscope compared to thin bronchoscope without fluoroscopy for peripheral pulmonary lesions. J Thorac Dis. 2022 May;14(5):1663-1673. doi: 10.21037/jtd-22-20. PMID 35693609